CLINICAL TRIAL: NCT04054193
Title: A Phase 4, Open-label, Single Arm Study to Evaluate the Safety and Tolerability of a Three-day Fosaprepitant Regimen Administered for the Prevention of Chemotherapy-Induced Nausea and Vomiting (CINV) in Pediatric Participants Receiving Emetogenic Chemotherapy
Brief Title: Safety of a Three-Day Fosaprepitant Regimen for the Prevention of Chemotherapy-Induced Nausea and Vomiting in Pediatric Participants (MK-0517-045)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0517-045; MK-0517-045 (Other: Merck); 2018-004844-43 (EudraCT Number)
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Results first posted 2021-09-23 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — fosaprepitant; Aprepitant; Serotonin 5-HT3 Receptor Antagonists; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fosaprepitant Treatment (Experimental): Participants received fosaprepitant dimeglumine once daily (QD) for 3 days and were followed for 14 days during the 17-day Cycle 1. Participants also optionally received dexamethasone as background therapy, and a serotonin (5-hydroxytryptamine [5-HT3]) receptor antagonist on Day 1 and optionally on Days 2-3 as background therapy. After completing Cycle 1, participants had the option to continue for up to 2 additional 17-day cycles of the same treatment regimen.
  Interventions: Drug: Fosaprepitant Dimeglumine; Drug: 5-HT3 antagonist; Drug: Dexamethasone

INTERVENTIONS:
Drug: Fosaprepitant Dimeglumine — Participants received IV fosaprepitant dimeglumine ≤115 mg on Day 1 and ≤80 mg on Days 2 and 3 (dose adjusted for age).
  Other Names: EMEND for injection®; MK-0517
Drug: 5-HT3 antagonist — All participants received an oral 5-hydroxytryptamine (serotonin; [5-HT]) 3 receptor antagonist on Day 1 and had the option to take on Days 2-3. The dose was as per product label or standard of care.
Drug: Dexamethasone — Participants received optional oral dexamethasone at the investigator's discretion according to product label or standard of care.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a 3-day intravenous (IV) fosaprepitant dimeglumine (MK-0517) regimen for the prevention of CINV in pediatric participants scheduled to receive emetogenic chemotherapy. Each participant was enrolled in Cycle 1 (on which the primary study objectives were based), consisting of the 3-day treatment cycle and 14 days of follow-up for a total of 17 days.

DETAILED DESCRIPTION:
Upon completion of Cycle 1, participants were given the option to exit the study and be considered completed, or to continue on study therapy for up to 2 more (optional) 17-day cycles of chemotherapy where fosaprepitant was administered and additional safety data collected.

ELIGIBILITY:
Inclusion Criteria:

* Is receiving a moderately or highly emetogenic chemotherapy agent/regimen or a chemotherapy agent/regimen not previously tolerated due to vomiting
* Has a Lansky Play Performance score ≥60 (participants ≤16 years of age) or a Karnofsky score ≥60 (participants >16 years of age)
* Has a pre-existing functional central venous catheter available for study treatment administration
* Is fosaprepitant naïve
* Has a predicted life expectancy ≥3 months
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: is not a woman of childbearing potential (WOCBP) OR is a WOCBP and agrees to not be sexually active or use a highly effective contraceptive method for at least 28 days prior to receiving study treatment, during the treatment period, and for at least 30 days (or local standard of care if longer) after the last dose of study treatment (including the optional cycles)
* Has a negative highly sensitive pregnancy test (urine or serum as required by local regulations) prior to the start of fosaprepitant administration in a given cycle if a WOCBP
* Weighs at least 6 kilograms (kg)

Exclusion Criteria:

* Will receive stem cell rescue therapy in conjunction with a study-related course of emetogenic chemotherapy or during the 14 days following administration of fosaprepitant
* Is currently a user of any recreational or illicit drugs or has current evidence of drug or alcohol abuse or dependence as determined by the investigator
* Is mentally incapacitated or has a significant emotional or psychiatric disorder that, in the opinion of the investigator, precludes study entry
* Is pregnant or breast feeding
* Is allergic to fosaprepitant, aprepitant, or prescribed 5-HT3 antagonist
* Has an active infection (eg, pneumonia), congestive heart failure, bradyarrhythmia, any uncontrolled disease (eg, diabetic ketoacidosis, gastrointestinal obstruction) except for malignancy, or has any illness which in the opinion of the investigator, might confound the results of the study or pose unwarranted risk in administering study treatment or concomitant therapy to the participant
* Is a WOCBP who has a positive pregnancy test at screening (Cycle 1) or on Day 1 of optional Cycles 2 or 3
* Has been started on systemic corticosteroid therapy within 72 hours prior to study treatment administration or is expected to receive a corticosteroid as part of the chemotherapy regimen. Exceptions apply
* Is taking excluded medications
* Has ever participated in a previous study of aprepitant or fosaprepitant or has taken a non-approved (investigational) drug within the last 4 weeks
* Has a known history of QT prolongation or is taking any medication that is known to lead to QT prolongation

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (26):
- United States (5):
  - Phoenix Childrens Hospital ( Site 1101), Phoenix, Arizona
  - Southern California Permanente Medical Group ( Site 1104), Los Angeles, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago ( Site 1106), Chicago, Illinois
  - Children's Hospitals and Clinics of Minnesota ( Site 1109), Minneapolis, Minnesota
  - St. Jude Children's Research Hospital ( Site 1111), Memphis, Tennessee
- Greece (3):
  - Athens Childrens Hospital Aglaia Kyriakou ( Site 0101), Athens, Attica
  - University of Athens - Aghia Sophia Childrens Hospital ( Site 0102), Athens, Attica
  - University General Hospital of Thessaloniki "AHEPA" ( Site 0103), Thessaloniki
- Hungary (3):
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi OktatoKorhaz ( Site 0203), Miskolc, Borsod-Abauj Zemplen county
  - Szegedi Tudomanyegyetem - Szent-Gyorgyi Albert Klinikai Kozpont ( Site 0201), Szeged, Csongrád megye
  - Heim Pal Orszagos Gyermekgyogyaszati Intezet ( Site 0202), Budapest
- Lithuania (2):
  - LSMUL Kauno Klinikos ( Site 0402), Kaunas
  - Vaiku ligonine VsI VUL Santaros kliniku filialas ( Site 0401), Vilnius
- Prinses Maxima Centrum ( Site 0501), Utrecht, Netherlands
- Peru (3):
  - Instituto Nacional de Enfermedades Neoplasicas ( Site 1502), Lima
  - Clinica Anglo Americana ( Site 1501), Lima
  - Clinica Delgado ( Site 1503), Lima
- Poland (2):
  - Instytut Matki i Dziecka ( Site 0601), Warsaw, Masovian Voivodeship
  - Instytut Pomnik Centrum Zdrowia Dziecka ( Site 0602), Warsaw, Masovian Voivodeship
- Russia (4):
  - Chelyabinsk Regional Children Clinical Hospital ( Site 0705), Chelyabinsk, Chelyabinsk Oblast
  - Blokhin National Medical Oncology ( Site 0701), Moscow, Moscow
  - Dmitry Rogachev National Research Center ( Site 0704), Moscow, Moscow
  - Clinical Research Center of specialized types medical care-Oncology ( Site 0706), Saint Petersburg, Sankt-Peterburg
- United Kingdom (3):
  - Leeds Teaching Hospitals NHS Trust ( Site 1002), Leeds
  - Alder Hey Childrens NHS Foundation Trust Hospital ( Site 1003), Liverpool
  - Royal Manchester Children's Hospital ( Site 1005), Manchester

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Garcia Leon JL, DiCristina C, Yao R, Afzal AS. Safety and Tolerability of a 3-Day Fosaprepitant Regimen for the Prevention of Chemotherapy-Induced Nausea and Vomiting in Pediatric Patients: Results of an Open-Label, Single-Arm Phase 4 Trial. Pediatr Hematol Oncol. 2025 Mar;42(2):79-91. doi: 10.1080/08880018.2024.2437047. Epub 2024 Dec 10. PMID 39655741
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were recruited at 25 study sites in 9 countries.
Groups:
- Fosaprepitant Treatment: Participants received fosaprepitant dimeglumine once daily (QD) for 3 days and were followed for 14 days during the 17-day Cycle 1. Participants also optionally received dexamethasone as background therapy, and a serotonin (5-hydroxytryptamine [5-HT]) 3 receptor antagonist on Day 1 and optionally on Days 2-3 as background therapy. After completing Cycle 1, participants had the option to continue for up to 2 additional 17-day cycles of the same treatment regimen.
Period: Cycle 1
Arm/Group | Fosaprepitant Treatment
Started | 103
Treated (≥1 Dose) | 100
Completed | 98
Not Completed | 5
Not completed — Physician Decision | 1
Not completed — Consent withdrawn by parent/guardian | 1
Not completed — Allocated but not treated | 3
Period: Cycles 2-3
Arm/Group | Fosaprepitant Treatment
Started | 69 (Participation in Cycles 2-3 was optional after completing Cycle 1.)
Completed (Completed Cycles 2 and 3) | 48
Not Completed | 21
Not completed — Physician Decision | 2
Not completed — Consent withdrawn by parent/guardian | 2
Not completed — Various reasons | 17

BASELINE CHARACTERISTICS:
Arm/Group | Fosaprepitant Treatment
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.7 (5.0) [lower limit 5.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 77
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 81
  More than one race | 6
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Cycle 1 Who Experienced One or More Adverse Events (AEs)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not it is considered related to the study drug. The percentage of participants in Cycle 1 who experience one or more AE(s) is presented.
Time Frame: Up to 17 days
Population: The analysis population consists of all allocated participants in Cycle 1 who received ≥1 dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant Treatment
Number analyzed (Participants) | 100
Percentage of Participants | 80.0

2. Primary Outcome: Percentage of Participants in Cycle 1 Who Discontinued Study Drug Due to an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not it is considered related to the study drug. The percentage of participants in Cycle 1 who discontinue study treatment due to an AE is presented.
Time Frame: Up to 3 days
Population: The analysis population consists of all allocated participants in Cycle 1 who received ≥1 dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant Treatment
Number analyzed (Participants) | 100
Percentage of Participants | 2.0

ADVERSE EVENTS:
Time Frame: Up to approximately 3.5 months
Description: All-cause mortality is reported for all allocated participants, and serious and nonserious adverse events are reported for all allocated participants who received ≥1 dose of study intervention. Findings from Cycle 1 and Cycles 2-3 are presented separately.
Groups:
- Fosaprepitant Cycle 1: Participants received fosaprepitant dimeglumine once daily (QD) for 3 days and were followed for 14 days during the 17-day Cycle 1. Participants also optionally received dexamethasone as background therapy, and a serotonin (5-hydroxytryptamine [5-HT]) 3 receptor antagonist on Day 1 and optionally on Days 2-3 as background therapy.
- Fosaprepitant Cycles 2-3: Participants received fosaprepitant dimeglumine once daily (QD) for 3 days and were followed for 14 days during Cycles 2-3. Participants also optionally received dexamethasone as background therapy, and a 5-HT3 receptor antagonist on Day 1 and optionally on Days 2-3 as background therapy, of each 17-day cycle.
Arm/Group | Fosaprepitant Cycle 1 | Fosaprepitant Cycles 2-3
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/69
Serious Adverse Events (participants affected / at risk) | 30/100 | 27/69
Other Adverse Events (participants affected / at risk) | 64/100 | 27/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant Cycle 1 (N=100) | Fosaprepitant Cycles 2-3 (N=69)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 4 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 17 (18) | 15 (20)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coordination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematotoxicity (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant Cycle 1 (N=100) | Fosaprepitant Cycles 2-3 (N=69)
Anaemia (Blood and lymphatic system disorders) | 24 (28) | 7 (8)
Haematotoxicity (Blood and lymphatic system disorders) | 9 (9) | 10 (15)
Neutropenia (Blood and lymphatic system disorders) | 15 (16) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (11) | 3 (3)
Constipation (Gastrointestinal disorders) | 6 (6) | 3 (3)
Nausea (Gastrointestinal disorders) | 24 (25) | 8 (9)
Vomiting (Gastrointestinal disorders) | 16 (18) | 8 (13)
Neutrophil count decreased (Investigations) | 14 (14) | 2 (2)
Platelet count decreased (Investigations) | 9 (9) | 4 (4)
White blood cell count decreased (Investigations) | 7 (8) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT04054193/Prot_SAP_001.pdf